CLINICAL TRIAL: NCT05830851
Title: Transcranial Direct Current Stimulation Combined With Aerobic Exercise for the Treatment of Chronic Nonspecific Low Back Pain: a Randomized Clinical Trial
Brief Title: Transcranial Direct Current Stimulation (tDCS) Combined With Aerobic Exercise in Chronic Nonspecific Low Back Pain (LBP)
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Marina Castel Sánchez, PhD, Physical Therapist and associated lecturer, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS&aeorbic excercise in LBP
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Low Back Pain; Chronic Low-back Pain
Keywords: low back pain; chronic low back pain; non-specific chronic low back pain; transcranial direct current stimulation; tDCS; aerobic exercise; aerobic training; walking
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aerobic exercise (Active Comparator): Walk on a treadmill during 20-30 minutes at 60-80% of Heart Rate max
  Interventions: Other: real tDCS and aerobic exercise; Other: sham tDCS and aerobic exercise
- Sham tDCS (Sham Comparator): Application of tDCS during 30 seconds of 2 mA-intensity.
  Interventions: Other: sham tDCS and aerobic exercise
- real tDCS (Experimental): Application of real tDCS during 20 minutes at 2 mili Amper (mA)-intensity.
  Interventions: Other: real tDCS and aerobic exercise

INTERVENTIONS:
Other: real tDCS and aerobic exercise — Walking on a treadmill at 60-80% of HRmax while wearing a head tDCS device with therapeutic parameters
  Arms: aerobic exercise; real tDCS
Other: sham tDCS and aerobic exercise — Walking on a treadmill at 60-80% of HRmax while wearing a head tDCS device with sham tDCS
  Arms: Sham tDCS; aerobic exercise

SUMMARY:
The goal of this clinical trial is to learn about the effects of transcranial direct current stimulation (tDCS) combined with aerobic exercise in non-specific low back pain patients. The main question aims to answer: • Which are the effects of tDCS treatment combined with aerobic exercise compared to Sham tDCS combined with aerobic exercise in non-specific Low Back Pain? Participants will be asked to complete questionnaires and they will receive treatments as tDCS or Sham tDCS and aerobic exercise (treadmill walking). Researchers will compare a group who is treated with a combination of tDCS and aerobic exercise versus a group receiving placebo tDCS and aerobic exercise to see the effects on pain intensity, pressure pain, disability, kinesiophobia, quality of life, catastrophism, Heart Rate Variability and cortical excitation.

DETAILED DESCRIPTION:
Low back pain (LBP) is the main cause of disability worldwide with a prevalence of 70 to 85% of the population. Chronic LBP (CLBP) is defined as a pain lasting more than 12 weeks. CLBP does not have peripheral nociceptive stimuli, but it is characterized by the presence of a chronic change in neuroplasticity. Transcranial direct current stimulation (tDCS) is a type of therapeutic intervention that can modulate the cortical excitability of a wide neural network involved in the elaboration of pain, resulting in an efficacy option for CLBP treatment. Aerobic exercise represents another typology of effective therapeutic intervention in the treatment of pain intensity and disability related to CLBP.

The main objective of the study is to determine the efficacy of tDCS combined with aerobic exercise compared to shame/placebo tDCS combined with aerobic exercise in middle-aged subjects with non-specific CLBP in the short, medium and long term.

Methods: In a double-blinded pilot randomized controlled trial, 38 subjects aged between 18 and 65 years, with a diagnose of non-specific LBP for 3 months, a Visual Analogue Scale (VAS) result of >20mm and a Roland-Morris Scale result of >4 will be selected for the following study. Participants will be divided in two groups of 19 subjects each one: experimental group A (20 minutes of tDCS at 2 mili Amper + 20-30 minutes of aerobic exercise at 60-80% of HRmax) and controlled group B (30 seconds of sham/placebo tDCS at 2milli amperes + 20-30 minutes of aerobic exercise at 60-80% of maximum heart rate). The following outcomes will be measured: pain intensity (100mm VAS), pressure pain (pressure algometer), disability (Roland-Morris questionnaire), kinesiophobia (Tampa Scale for kinesiophobia), quality of life (SF-12 health questionnaire), catastrophism (Pain Catastrophizing Scale), Heart Rate Variability ( Polar Team) and cortical excitation (Critical Flicker Fusion).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-specific Low Back Pain for at least 3 months based on careful radiological evaluation and clinical diagnosis by a physician.
* Aged from 18 till 65 years old.
* Scoring higher than 20mm on the 100 mm VAS scale
* Scoring higher than 4 on the Rolland-Morris scale

Exclusion Criteria:

Any subject presenting at least one of the following exclusion criteria will be excluded from the study:

* Vertebral fractures, osteoporosis
* Infections
* Lumbar surgical, herniated disc or nerve root compression
* Rheumatologic diseases
* People with central nervous system alterations
* Structured deformities of the spine (scoliosis)
* Oncology patients in active treatment or within 5 years after the end of the treatment
* Fibromyalgia
* Women who are pregnant or who may be pregnant
* Contraindications to tDCS (epilepsy, cranial implanted devices, neurological o psychiatric disorders, sever cardiopulmonary, renal or hepatic disorders)
* Being under physiotherapeutic or osteopathic treatment during the study period
* Absolute contraindications to aerobic exercise (acute myocardial infarction, unstable angina pectoris, uncontrolled arrhythmia, heart failure, acute pulmonary embolism, myocarditis or acute pericarditis)
* People who need walking assistance (cane, other person to assist)
* Patients who practise regular physical activity defined as leisure-time physical activity for 30 minutes, three or more times per week
* People unable to give informed consent, or unable to complete the selected questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-17 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At baseline
  Measured with Visual Analogue Scale of 100 mm
Pain intensity | At the first month after intervention onset (after completion of the 12 treatment sessions).
  Measured with Visual Analogue Scale of 100 mm
Pain intensity | Follow-up at the third month after treatment completion
  Measured with Visual Analogue Scale of 100 mm
Pain intensity | Follow-up at the sixth month after treatment completion
  Measured with Visual Analogue Scale of 100 mm
Pressure pain | At baseline
  Measured with a pressure algometer
Pressure pain | At the first month after intervention onset (after completion of the 12 treatment sessions).
  Measured with a pressure algometer
Pressure pain | Follow-up at the third month after treatment completion
  Measured with a pressure algometer
Pressure pain | Follow-up at the sixth month after treatment completion
  Measured with a pressure algometer

SECONDARY OUTCOMES:
Disability | At baseline
  Measured with Roland-Morris scale Spanish version, minimum and maximum values go from 0 (absence of disability) until 24 (maximum disability)
Disability | At the first month after intervention onset (after completion of the 12 treatment sessions).
  Measured with Roland-Morris scale Spanish version, minimum and maximum values go from 0 (absence of disability) until 24 (maximum disability)
Disability | Follow-up at the third month after treatment completion
  Measured with Roland-Morris scale Spanish version, minimum and maximum values go from 0 (absence of disability) until 24 (maximum disability)
Disability | Follow-up at the sixth month after treatment completion
  Measured with Roland-Morris scale Spanish version, minimum and maximum values go from 0 (absence of disability) until 24 (maximum disability)
Kinesiophobia | At baseline
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Kinesiophobia | At the first month after intervention onset (after completion of the 12 treatment sessions)
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Kinesiophobia | Follow-up at the third month after treatment completion
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Kinesiophobia | Follow-up at the sixth month after treatment completion
  Measured with Tampa Kinesiophobia Scale questionnaire (TSK-11SV) Spanish version. Minimum and maximum values are between 11 and 44 point, a result with higher values indicates higher level of kinesiofobia.
Quality of life questionnaire | Al baseline
  Measured with SF-12 Health Questionnaire Spanish version. A zero score indicates the lowest level of dimension measured by the scale, and 100 indicates the highest level of the measured dimension
Quality of life questionnaire | At the first month after intervention onset (after completion of the 12 treatment sessions)
  Measured with SF-12 Health Questionnaire Spanish version. A zero score indicates the lowest level of dimension measured by the scale, and 100 indicates the highest level of the measured dimension
Quality of life questionnaire | Follow-up at the third month after treatment completion
  Measured with SF-12 Health Questionnaire Spanish version. A zero score indicates the lowest level of dimension measured by the scale, and 100 indicates the highest level of the measured dimension
Quality of life questionnaire | Follow-up at the sixth month after treatment completion
  Measured with SF-12 Health Questionnaire Spanish version. A zero score indicates the lowest level of dimension measured by the scale, and 100 indicates the highest level of the measured dimension
Catastrophism | At baseline
  Measured with Pain Catastrophism Scale Spanish version. The total score ranges from 0 to 52. Higher scores reflect higher levels of catastrophic thinking.
Catastrophism | At the first month after intervention onset (after completion of the 12 treatment sessions)
  Measured with Pain Catastrophism Scale Spanish version. The total score ranges from 0 to 52. Higher scores reflect higher levels of catastrophic thinking.
Catastrophism | Follow-up at the third month after treatment completion
  Measured with Pain Catastrophism Scale Spanish version. The total score ranges from 0 to 52. Higher scores reflect higher levels of catastrophic thinking.
Catastrophism | Follow-up at the sixth month after treatment completion
  Measured with Pain Catastrophism Scale Spanish version. The total score ranges from 0 to 52. Higher scores reflect higher levels of catastrophic thinking.
Cortical excitation | At baseline
  Measured with Critical Flicker Fusion Threshold
Cortical excitation | At the first month after intervention onset (after completion of the 12 treatment sessions)
  Measured with Critical Flicker Fusion Threshold
Cortical excitation | Follow-up at the third month after treatment completion
  Measured with Critical Flicker Fusion Threshold
Cortical excitation | Follow-up at the sixth month after treatment completion
  Measured with Critical Flicker Fusion Threshold
Heart Rate Variability | At baseline
  Measured with Polar Heart Rate belt
Heart Rate Variability | At the first month after intervention onset (after completion of the 12 treatment sessions)
  Measured with Polar Heart Rate belt
Heart Rate Variability | Follow-up at the third month after treatment completion
  Measured with Polar Heart Rate belt
Heart Rate Variability | Follow-up at the sixth month after treatment completion
  Measured with Polar Heart Rate belt

CONTACTS AND LOCATIONS:
Overall Officials: Marina Castel Sánchez, PhD, Principal Investigator — European University of Madrid.Department of Physiotherapy, Chiropody and Dance
Locations (2):
- Spain (2):
  - Eurpean University of Madrid, Villaviciosa de Odón, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alwardat M, Pisani A, Etoom M, Carpenedo R, Chine E, Dauri M, Leonardis F, Natoli S. Is transcranial direct current stimulation (tDCS) effective for chronic low back pain? A systematic review and meta-analysis. J Neural Transm (Vienna). 2020 Sep;127(9):1257-1270. doi: 10.1007/s00702-020-02223-w. Epub 2020 Jul 9. PMID 32647923
- [Background] Wong CK, Mak RY, Kwok TS, Tsang JS, Leung MY, Funabashi M, Macedo LG, Dennett L, Wong AY. Prevalence, Incidence, and Factors Associated With Non-Specific Chronic Low Back Pain in Community-Dwelling Older Adults Aged 60 Years and Older: A Systematic Review and Meta-Analysis. J Pain. 2022 Apr;23(4):509-534. doi: 10.1016/j.jpain.2021.07.012. Epub 2021 Aug 24. PMID 34450274
- [Background] Pergolizzi JV Jr, LeQuang JA. Rehabilitation for Low Back Pain: A Narrative Review for Managing Pain and Improving Function in Acute and Chronic Conditions. Pain Ther. 2020 Jun;9(1):83-96. doi: 10.1007/s40122-020-00149-5. Epub 2020 Jan 31. PMID 32006236
- [Background] Tornero Aguilera JF, Fernandez Elias V, Clemente-Suarez VJ. Autonomic and cortical response of soldiers in different combat scenarios. BMJ Mil Health. 2021 Jun;167(3):172-176. doi: 10.1136/jramc-2019-001285. Epub 2020 Feb 27. PMID 32111675
- [Background] Cavalcante PGL, Baptista AF, Cardoso VS, Filgueiras MC, Hasue RH, Joao SMA, Hazime FA. Transcranial Direct Current Stimulation Combined With Therapeutic Exercise in Chronic Low Back Pain: Protocol of a Randomized Controlled Trial. Phys Ther. 2020 Aug 31;100(9):1595-1602. doi: 10.1093/ptj/pzaa105. PMID 32526017
- [Background] Ouellette AL, Liston MB, Chang WJ, Walton DM, Wand BM, Schabrun SM. Safety and feasibility of transcranial direct current stimulation (tDCS) combined with sensorimotor retraining in chronic low back pain: a protocol for a pilot randomised controlled trial. BMJ Open. 2017 Aug 21;7(8):e013080. doi: 10.1136/bmjopen-2016-013080. PMID 28827229
- [Background] Pinto CB, Teixeira Costa B, Duarte D, Fregni F. Transcranial Direct Current Stimulation as a Therapeutic Tool for Chronic Pain. J ECT. 2018 Sep;34(3):e36-e50. doi: 10.1097/YCT.0000000000000518. PMID 29952860
- [Background] DosSantos MF, Ferreira N, Toback RL, Carvalho AC, DaSilva AF. Potential Mechanisms Supporting the Value of Motor Cortex Stimulation to Treat Chronic Pain Syndromes. Front Neurosci. 2016 Feb 11;10:18. doi: 10.3389/fnins.2016.00018. eCollection 2016. PMID 26903788
- [Background] Pacheco-Barrios K, Cardenas-Rojas A, Thibaut A, Costa B, Ferreira I, Caumo W, Fregni F. Methods and strategies of tDCS for the treatment of pain: current status and future directions. Expert Rev Med Devices. 2020 Sep;17(9):879-898. doi: 10.1080/17434440.2020.1816168. Epub 2020 Sep 15. PMID 32845195
- [Background] Bruehl S, Burns JW, Koltyn K, Gupta R, Buvanendran A, Edwards D, Chont M, Wu YH, Qu'd D, Stone A. Are endogenous opioid mechanisms involved in the effects of aerobic exercise training on chronic low back pain? A randomized controlled trial. Pain. 2020 Dec;161(12):2887-2897. doi: 10.1097/j.pain.0000000000001969. PMID 32569082
- [Background] O'Connor SR, Tully MA, Ryan B, Bleakley CM, Baxter GD, Bradley JM, McDonough SM. Walking exercise for chronic musculoskeletal pain: systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 Apr;96(4):724-734.e3. doi: 10.1016/j.apmr.2014.12.003. Epub 2014 Dec 19. PMID 25529265